CLINICAL TRIAL: NCT05873803
Title: A Randomized, Double Blind, Placebo-Controlled Phase II Study to Evaluate the Efficacy, Safety of GR1802 Injection in Patients with Chronic Rhinosinusitis with Nasal Polyps (CRSwNP)
Brief Title: The Study of GR1802 in Patients with Chronic Rhinosinusitis with Nasal Polyps
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Genrix (Shanghai) Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GR1802-005
Record Dates: First submitted 2023-05-16; First posted 2023-05-24 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-06

CONDITIONS: Chronic Rhinosinusitis with Nasal Polyps

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: GR1802 (Experimental): GR1802 injection 300mg every two weeks for 16-week treatment
  Interventions: Biological: GR1802 injection
- Placebo Comparator: Placebo (Placebo Comparator): Placebo every two weeks for 16-week treatment
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: GR1802 injection — 150mg/1ml. 2 ml every two weeks Route of administration: Subcutaneous
  Arms: Experimental: GR1802
Biological: placebo — 0mg/1ml. 2 ml every two weeks Route of administration: Subcutaneous
  Arms: Placebo Comparator: Placebo

SUMMARY:
This is a multi-center, randomized, double blind, placebo-controlled study to evaluate the efficacy, safety, PK, PD and immumogenicity of GR1802 injection in comparison to placebo in addition to a background treatment of mometasone furcate nasal spray (MFNS) in patients with chronic rhinosinusitis with nasal polyposis (CRSwNP). Patients will receive GR1802 injection or Placebo every 2 Weeks.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled phase II clinical trial evaluating the preliminary efficacy and safety of GR1802 injection in patients with chronic rhinosinusitis with nasal polyps.

The study consists of a Screening/run-in Period (up to 4 weeks), a Randomized, Double Blind Treatment Period (16 weeks) and a Safety Follow-up Period (8 weeks).

70 subjects will be randomized 1:1 into the 300 mg first dose doubling Q2W group and the placebo Q2W group. Throughout the dosing period, all subjects continued treatment with standard therapy at a stable dose.

Patient-reported outcome including Nasal congestion score will be collected using patient diary. Central reading will be implemented to Nasal endoscopic nasal polyp score (NPS) and nasal polyp biopsy tissue analysis to eosinophil counts & percentage.

ELIGIBILITY:
Inclusion Criteria:

1. Bilateral CRSwNP with prior treatment with systemic corticosteroids (SCS), and/or contraindicate to or intolerance to SCS, and/or with prior surgery to nasal polyps
2. Bilateral NPS of ≥5 with a minimum score of 2 in each nasal cavity at screening and at baseline.
3. Ongoing symptoms of nasal congestion/obstruction(NCS score of 2 or 3 at screening and at baseline).
4. Recorded use of intranasal corticosteroids for at least 4 weeks before screening

Exclusion Criteria:

1. Insufficient washout time for drugs that have an impact on the evaluation of efficacy and safety。
2. Concurrent disease that may interfere with the evaluation of safety and efficacy in subjects, or affect the risk- benefit evaluation of subjects. eg. specific ongoing nasal diseases, severe asthma, active infection, Severe cardiovascular disease, Severe laboratory test abnormalities.
3. Other.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-02-08 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline at Week 16 in Nasal Congestion/Obstruction Symptom(NCS) Severity Score | at Week 16
  Change from baseline in the NCS score. NCS score (0-3), higher score means worse nasal symptom.
Change From Baseline at Week 16 in Nasal Polyp Score | at Week 16
  NPS score ranges from 0-8. (sum of 0-4 for each nasal passage scores), higher score means a worse outcome.

SECONDARY OUTCOMES:
Time to the first response of NPS | Baseline up to Week 24
  Time to the first response of NPS (defined as bilateral endoscopic NPS improved ≥1).
Lund-Mackay score | at Week 16
  Change from baseline in the Lund-Mackay score on CT scan. The range of LM score is 0-24. Higher score means worse rhinosinusitis.
Bilateral endoscopic NPS | at Week 4, 8, 12, 24
  Change from baseline in the bilateral endoscopic NPS at Week 4, 8, 12, 24.
Nasal Congestion/Obstruction Symptom score(NCS) | at Week 4, 8, 12, 24
  Change from baseline in NCS at Week 4, 8, 12, 24.
University of Pennsylvania Smell Identification Test (UPSIT) | at Week 16
  Change from baseline in UPSIT. UPSIT score (0-40). Higher score means better sense of smell.
Total Nasal Symptom Score(TNSS) score | at Week 16
  Change from baseline in TNSS score. TNSS score (0-9). Higher score means worse nasal symptom.
Visual Analogue Scale (VAS) for Rhinosinusitis | at Week 16
  Change from baseline in VAS score. VAS score (0-10). Higher score means worse nasal symptom.
Proportion of subjects receiving rescue therapy for nasal polyps | Baseline up to Week 24
  Rescue therapy includes Systemic Corticosteroids and endoscopic surgery
Pharmacokinetics(PK) | Baseline up to Week 24
  Plasma concentration of GR1802 injection. PK parameter including trough concentration and exposure（CL/F, Vz/F etc.）
Pharmacodynamics(PD) | at Week 16
  Change from baseline in serum biomarker level (Periostin, TARC, total IgE and eosinophil level) and biomarkers in nasal secretions and nasal exfoliated cells。
Anti-drug antibodies(ADA) | Baseline up to Week 24
  Incidence of ADA
Safety parameters | Baseline up to Week 24
  Incidence of treatment-emergent adverse events (TEAEs), of treatment-emergent serious AEs (TESAEs), etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No